CLINICAL TRIAL: NCT04295135
Title: Nudging Primary Care Providers Toward Guideline-Recommended Opioid Prescribing Through Easier and More Convenient EHR Information Design
Brief Title: Chronic Pain OneSheet Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Eskenazi Health (Other); Wake Forest University (Other); Wake Forest University Health Sciences (Other); University of Florida (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Olena Mazurenko, Principal Investigator, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1911922583; 5R33DA046085-05 (NIH)
Record Dates: First submitted 2020-02-15; First posted 2020-03-04 (Actual); Results first posted 2024-05-24 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Chronic Pain
Keywords: Clinical Decision Support; Chronic pain care; Behavioral Economics; Provider behavior
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OneSheet access (Experimental): PCPs who receive access to, and training in the Chronic Pain OneSheet, and use it while caring for patients with chronic pain.
  Interventions: Behavioral: Chronic Pain OneSheet
- Normal practice (No Intervention): PCPs who do not receive access to, or training in the Chronic Pain OneSheet, and care for patients with chronic pain as they would normally.

INTERVENTIONS:
Behavioral: Chronic Pain OneSheet — The Chronic Pain OneSheet (OneSheet) is an EHR decision support tool that uses behavioral economics to increase adoption of chronic pain guideline recommendations. OneSheet works by aggregating and structuring information that is already collected, that PCPs often need while caring for patients with chronic pain conditions. By aggregating and structuring this information in a more convenient manner, the goal of OneSheet is to make the information that is important in clinical decision making more readily available, and to reduce the amount of time that PCPs need to spend locating this information.
  Other Names: Pain Dashboard
  Arms: OneSheet access

SUMMARY:
The purpose of the study is to determine whether and how having access to the Chronic Pain OneSheet clinical decision support tool in Epic affects the ordering, prescribing, goal-setting, risk monitoring, and outcome measuring behavior of participating primary care providers (PCPs) in visits with patients with chronic pain conditions. The investigators will also assess whether access to the Chronic Pain OneSheet results in PCPs making chronic pain treatment decisions that are more concordant with the Centers for Disease Control and Prevention (CDC) Guideline for Prescribing Opioids for Chronic Pain.

DETAILED DESCRIPTION:
The Chronic Pain OneSheet (OneSheet) is an electronic health record (EHR) based clinical support tool developed and built in Epic. The OneSheet is a dashboard designed to assist PCPs in treating patients with chronic pain conditions by providing an overview of patient information needed by PCPs when treating these patients. The dashboard does not provide new information to PCPs. Instead, it works by aggregating and structuring information already being collected, available in other places in the medical record. By aggregating and structuring this information more conveniently, the goal of the OneSheet is to make important information in clinical decision-making more readily available and reduce the time PCPs need to spend locating this information.

The study aimed to determine whether and how having access to the Chronic Pain OneSheet activity in Epic affects the ordering, prescribing, goal-setting, risk monitoring, and outcome-measuring behavior of participating PCPs in visits with patients with chronic pain conditions. The investigators also assessed whether access to the Chronic Pain OneSheet results in PCPs making chronic pain treatment decisions that are more concordant with the CDC Guideline for Prescribing Opioids for Chronic Pain.

To test this, researchers conducted a two-arm pragmatic randomized controlled trial (RCT), enrolling PCPs across two health systems. The randomization occurred at the PCP level; the analysis occurred at the patient-visit level. The PCPs signed an informed consent form, while the data from patient visits was obtained through a waiver of informed consent. The investigators assessed outcomes by analyzing EHR usage log files and PCP ordering records extracted from the healthcare systems' clinical data warehouses.

ELIGIBILITY:
Inclusion Criteria:

* Primary care provider (including Family Medicine, Internal Medicine, Med-Peds, and General Medicine)
* Can prescribe medication (i.e., Doctor of Medicine (MD), Nurse Practitioner (NP), Physicians Assistant (PA))
* Sees patients at a primary care clinic at one of the two participating hospital systems

Exclusion Criteria:

* Does not practice primary care
* Does not regularly see patients at a primary care clinic at one of the two participating hospital systems
* Cannot prescribe medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2020-08-04 (Actual); Primary Completion 2022-05-18 (Actual); Study Completion 2022-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher A Harle, PhD, Principal Investigator — Indiana University; Olena Mazurenko, MD, PhD, Principal Investigator — Indiana University
Locations (2):
- United States (2):
  - Indiana University, Indianapolis, Indiana
  - Wake Forest University, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mazurenko O, Sanner L, Apathy NC, Mamlin BW, Menachemi N, Adams MCB, Hurley RW, Erazo SF, Harle CA. Evaluation of electronic recruitment efforts of primary care providers as research subjects during the COVID-19 pandemic. BMC Prim Care. 2022 Apr 28;23(1):95. doi: 10.1186/s12875-022-01705-y. PMID 35484491

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Primary care providers (PCP) were recruited after virtual staff meetings. PCP recruitment occurred in two phases: Phase 1(health system 1: Aug-Oct 2020; health system 2: Sept-Nov 2020) and Phase 2 (Sep-Dec 2021). Phase 2 recruited more PCPs to increase the sample size and allow new PCPs to participate. PCPs were randomly assigned to either a treatment or a control group (permanent assignment). We combined data from PCPs recruited in both phases for analysis.
Groups:
- OneSheet Access: PCPs who receive access to, and training in the Chronic Pain OneSheet, and use it while caring for patients with chronic pain.
  Chronic Pain OneSheet: The Chronic Pain OneSheet (OneSheet) is an electronic health record (EHR) decision support tool that uses behavioral economics to increase adoption of chronic pain guideline recommendations. OneSheet works by aggregating and structuring information that is already collected, that PCPs often need while caring for patients with chronic pain conditions. By aggregating and structuring this information in a more convenient manner, the goal of OneSheet is to make the information that is important in clinical decision making more readily available, and to reduce the amount of time that PCPs need to spend locating this information.
Period: Overall Study
Arm/Group | OneSheet Access | Normal Practice
Started | 69 (64 PCPs were enrolled in the OneSheet Access group during recruitment phase #1. 5 PCPs were added in recruitment phase #2) | 68 (63 PCPs were enrolled to the Normal Practice group during recruitment phase #1. 5 PCPs were added in recruitment phase #2.)
Completed | 59 | 63
Not Completed | 10 | 5
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Subject left organization | 8 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OneSheet Access | Normal Practice | Total
Number analyzed (Participants) | 69 | 68 | 137
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 68 | 68 | 136
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 40 | 88
  Male | 21 | 28 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 8 | 12
  Not Hispanic or Latino | 54 | 47 | 101
  Unknown or Not Reported | 11 | 13 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 7 | 2 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 6 | 10
  White | 52 | 52 | 104
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 5 | 8 | 13
Region of Enrollment [Number; unit: participants]
  United States | 69 | 68 | 137
Years practicing medicine [Mean (Standard Deviation); unit: years] | 10.2 (9.94) | 9.7 (9.39) | 10.0 (9.64)

OUTCOME MEASURES:

1. Primary Outcome: Pain and Function Goal-setting
Description: Proportion of visits for patients with chronic pain for whom the PCP documented pain and/or function goals in the EHR, as assessed by data extracted from the healthcare systems' clinical data warehouse.
Time Frame: Assessed at baseline (looked back at previous 12 months) and 18-month treatment period
Population: PCPs enrolled during both recruitment phases and their visits with adult patients with chronic pain starting at the baseline (looked back at previous 12 months; pre-OneSheet Go-Live) and 18-month treatment period (post-OneSheet Go-Live).
Measure: Mean (Standard Deviation); unit: Proportion of patient visits
Units Other Than Participants: Patient visits
Arm/Group | OneSheet Access | Normal Practice
Number analyzed (Participants) | 69 | 66
Number analyzed (Patient visits) | 252625 | 220179
Proportion of patient visits
  Pre OneSheet Go-Live: number analyzed (Patient visits) | 107114 | 93111
  Pre OneSheet Go-Live | 0.0081 (0.0898) | 0.0016 (0.0404)
  Post OneSheet Go-Live: number analyzed (Patient visits) | 145511 | 127068
  Post OneSheet Go-Live | 0.0364 (0.1873) | 0.0283 (0.1659)
Statistical Analysis 1: Comparison: OneSheet Access vs Normal Practice; Test type: Superiority; p < 0.05, Regression, Linear — A multi-level linear probability model that included patient demographics, clinician random effects, and indicator variables for (a) site; (b) treatment and control clinicians; and (c) pre-/post-OneSheet access; Model also included an interaction term for treatment and post-OneSheet access; Mean Difference (Net) = 0.002, Standard Error of Mean 0.001 — The coefficient estimates the causal effect of OneSheet on our outcomes. Unit of analysis was patient visit

2. Primary Outcome: Pain, Enjoyment of Life, and General Activity (PEG) Documentation
Description: Proportion of visits for patients with chronic pain for whom the PCP documented the assessment of pain and/or function (e.g. Pain, Enjoyment, General Activity (PEG) scale in the EHR, as assessed by data extracted from the healthcare systems' clinical data warehouse. The PEG has a scale of 1-10, and is used to track an individual's changes over time. With effective therapy, an individual's score should decrease over time.
Time Frame: Assessed at baseline (looked back at previous 12 months) and 18-month treatment period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Proportion of patient visits
Units Other Than Participants: Patient visits
Arm/Group | OneSheet Access | Normal Practice
Number analyzed (Participants) | 69 | 66
Number analyzed (Patient visits) | 252625 | 220179
Proportion of patient visits
  Pre OneSheet Go-Live: number analyzed (Patient visits) | 107114 | 93111
  Pre OneSheet Go-Live | 0.0086 (0.0923) | 0.0096 (0.0973)
  Post OneSheet Go-Live: number analyzed (Patient visits) | 145511 | 127068
  Post OneSheet Go-Live | 0.0313 (0.1741) | 0.0253 (0.1572)
Statistical Analysis 1: Comparison: OneSheet Access vs Normal Practice; Test type: Superiority; p < 0.01, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Model also included an interaction term for treatment and post-OneSheet access; Median Difference (Net) = 0.007, Standard Error of Mean 0.001 — The coefficient estimates the causal effect of OneSheet on our outcomes. Unit of analysis was patient visit

3. Primary Outcome: Urine Drug Screening (UDS) Results Ordered
Description: Proportion of visits for patients with chronic pain on long term opioid therapy (LTOT) for whom the PCP ordered a UDS, as assessed by data extracted from the healthcare systems' clinical data warehouse.
Time Frame: Assessed at baseline (looked back at previous 12 months) and 18-month treatment period
Population: PCPs enrolled during both recruitment phases and their visits with adult patients with chronic pain on LTOT starting at the baseline (looked back at previous 12 months; pre-OneSheet Go-Live) and 18-month treatment period (post-OneSheet Go-Live). The number of units (patient visits and participant counts) analyzed differs between the pre-OneSheet Go-Live and post-OneSheet Go-Live periods due to some PCPs only having qualifying visits in either the pre- or post- intervention period.
Measure: Mean (Standard Deviation); unit: Proportion of patient visits
Units Other Than Participants: Patient visits
Arm/Group | OneSheet Access | Normal Practice
Number analyzed (Participants) | 67 | 65
Number analyzed (Patient visits) | 26942 | 23492
Proportion of patient visits
  Pre OneSheet Go-Live: number analyzed (Participants) | 63 | 61
  Pre OneSheet Go-Live: number analyzed (Patient visits) | 11462 | 10492
  Pre OneSheet Go-Live | 0.4175 (0.4932) | 0.5486 (0.4977)
  Post OneSheet Go-Live: number analyzed (Participants) | 64 | 65
  Post OneSheet Go-Live: number analyzed (Patient visits) | 15480 | 13000
  Post OneSheet Go-Live | 0.3746 (0.4840) | 0.4705 (0.4991)
Statistical Analysis 1: Comparison: OneSheet Access vs Normal Practice; Test type: Superiority; p < 0.01, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Model also included an interaction term for treatment and post-OneSheet access; Mean Difference (Net) = 0.022, Standard Error of Mean 0.008 — The coefficient estimates the causal effect of OneSheet on our outcomes. Unit of analysis was patient visit

4. Primary Outcome: Prescription Drug Monitoring Program (PDMP) Reports Reviewed
Description: Proportion of visits for patients with chronic pain on LTOT for whom the PCP accessed the PDMP report, as assessed by data extracted from the healthcare systems' clinical data warehouse.
Time Frame: Assessed at baseline (looked back at previous 12 months) and 18-month treatment period
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Proportion of patient visits
Units Other Than Participants: Patient visits
Arm/Group | OneSheet Access | Normal Practice
Number analyzed (Participants) | 67 | 65
Number analyzed (Patient visits) | 26942 | 23492
Proportion of patient visits
  Pre OneSheet Go-Live: number analyzed (Participants) | 63 | 61
  Pre OneSheet Go-Live: number analyzed (Patient visits) | 11462 | 10492
  Pre OneSheet Go-Live | 0.7457 (0.4355) | 0.7962 (0.4028)
  Post OneSheet Go-Live: number analyzed (Participants) | 64 | 65
  Post OneSheet Go-Live: number analyzed (Patient visits) | 15480 | 13000
  Post OneSheet Go-Live | 0.8008 (0.3994) | 0.8461 (0.3609)
Statistical Analysis 1: Comparison: OneSheet Access vs Normal Practice; Test type: Superiority; p > 0.05, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Model also included an interaction term for treatment and post-OneSheet access; Median Difference (Net) = -0.005, Standard Error of Mean 0.006 — The coefficient estimates the causal effect of OneSheet on our outcomes. Unit of analysis was patient visit

5. Secondary Outcome: Naloxone Prescriptions Ordered
Description: Proportion of visits for patients with chronic pain on LTOT for whom the PCP ordered naloxone, as assessed by data extracted from the healthcare systems' clinical data warehouse.
Time Frame: Assessed at baseline (looked back at previous 12 months) and 18-month treatment period
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Proportion of patient visits
Units Other Than Participants: Patient visits
Arm/Group | OneSheet Access | Normal Practice
Number analyzed (Participants) | 67 | 65
Number analyzed (Patient visits) | 26942 | 23492
Proportion of patient visits
  Pre OneSheet Go-Live: number analyzed (Participants) | 63 | 61
  Pre OneSheet Go-Live: number analyzed (Patient visits) | 11462 | 10492
  Pre OneSheet Go-Live | 0.0012 (0.0349) | 0.0004 (0.0195)
  Post OneSheet Go-Live: number analyzed (Participants) | 64 | 65
  Post OneSheet Go-Live: number analyzed (Patient visits) | 15480 | 13000
  Post OneSheet Go-Live | 0.0054 (0.0730) | 0.0090 (0.0944)
Statistical Analysis 1: Comparison: OneSheet Access vs Normal Practice; Test type: Superiority; p < 0.01, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Model also included an interaction term for treatment and post-OneSheet access; Median Difference (Net) = -0.005, Standard Error of Mean 0.001 — The coefficient estimates the causal effect of OneSheet on our outcomes. Unit of analysis was patient visit

6. Secondary Outcome: Medications for Opioid Use Disorder Prescription Ordered
Description: Proportion of visits for patients with chronic pain on LTOT for whom the PCP ordered a medication for opioid use disorder, as assessed by data extracted from the healthcare systems' clinical data warehouse.
Time Frame: Assessed at baseline (looked back at previous 12 months) and 18-month treatment period
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Proportion of patient visits
Units Other Than Participants: Patient visits
Arm/Group | OneSheet Access | Normal Practice
Number analyzed (Participants) | 67 | 65
Number analyzed (Patient visits) | 26942 | 23492
Proportion of patient visits
  Pre OneSheet Go-Live: number analyzed (Participants) | 63 | 61
  Pre OneSheet Go-Live: number analyzed (Patient visits) | 11462 | 10492
  Pre OneSheet Go-Live | 0.0119 (0.1083) | 0.0092 (0.0957)
  Post OneSheet Go-Live: number analyzed (Participants) | 64 | 65
  Post OneSheet Go-Live: number analyzed (Patient visits) | 15480 | 13000
  Post OneSheet Go-Live | 0.0383 (0.1919) | 0.0373 (0.1895)
Statistical Analysis 1: Comparison: OneSheet Access vs Normal Practice; Test type: Superiority; p > 0.05, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Model also included an interaction term for treatment and post-OneSheet access; Median Difference (Net) = -0.002, Standard Error of Mean 0.003 — The coefficient estimates the causal effect of OneSheet on our outcomes. Unit of analysis was patient visit

ADVERSE EVENTS:
Time Frame: 18 month treatment period
Arm/Group | OneSheet Access | Normal Practice
All-Cause Mortality (participants affected / at risk) | 0/69 | 0/68
Serious Adverse Events (participants affected / at risk) | 0/69 | 0/68
Other Adverse Events (participants affected / at risk) | 0/69 | 0/68

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2024-01-09): https://cdn.clinicaltrials.gov/large-docs/35/NCT04295135/Prot_001.pdf
  • Statistical Analysis Plan (2024-03-05): https://cdn.clinicaltrials.gov/large-docs/35/NCT04295135/SAP_002.pdf
  • Informed Consent Form (2021-07-27): https://cdn.clinicaltrials.gov/large-docs/35/NCT04295135/ICF_003.pdf